CLINICAL TRIAL: NCT05429333
Title: Effect of Artificial Intelligence-assisted Personalized Microbiome Modulation by Diet in Functional Constipation: a Randomized Controlled Trial
Brief Title: Effect of Microbiome Modulation by Diet in Functional Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10840098-772.02-E.47859
Record Dates: First submitted 2022-06-17; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Constipation - Functional
Keywords: Microbiome; Artificial intelligence; Diet; Functional bowel disorders; Brain-gut diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): After randomization control group was recommended to continue their regular diet with increased fluid (2 lt/day) and fiber intake (30 g/day) and received 5 mg of sodium picosulfate daily for 10 weeks.
- Treatment group (Experimental): In the study group, after fecal samples were taken, patients were recommended to continue their regular diet with increased fluid (2 lt/day) and fiber intake (30 g/day) for 4 weeks until the microbiome analysis resulted. During subsequent 6 weeks, they received the personalized microbiome modulatory diet.
  Interventions: Other: Artificial intelligence-assisted personalized diet

INTERVENTIONS:
Other: Artificial intelligence-assisted personalized diet — The AI-based nutritional recommendations system is based on the eating rates of the individual in a certain period, to ensure the homeostasis of the microbiome and increase the microbial diversity.
  After the microbiome analysis reports of the study group are released, a 6-week diet was designed regarding AI-based food scores specific to constipated individuals in accordance with the individual's lifestyle and comorbidities. Diet lists are updated according to the individual's feedback, recovery level, and wishes with weekly meetings.
  Arms: Treatment group

SUMMARY:
Current medications and behavioral modifications have limited success in the treatment of functional constipation (FC). An individualized diet based on microbiome analysis may improve symptoms in FC. In the present study, we aimed to investigate the impacts of microbiome modulation on chronic constipation. patients fulfilling Rome IV criteria for functional constipation were randomized into two groups. The Control group received sodium picosulfate plus conventional treatments (i.e., laxatives, enemas, increased fiber, and fluid intake). The study group underwent microbiome analysis and received an individualized diet with the assistance of a soft computing system (Enbiosis Biotechnology®, Sariyer, Istanbul). Differences in Patient Assessment Constipation-Quality of Life (PAC-QoL) score and complete bowel movements per week (CBMpW) were compared between groups after 6 week-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilling Rome IV criteria for functional constipation (FC)
* Patients who had a colonoscopy performed within the last 5 years
* Patients who had a colonic transit time assessment within the last 3 months
* Patients who had a magnetic resonance defecography within the last 3 months

Exclusion Criteria:

* Use of antibiotics, probiotics, and/or prebiotics within the last 4 weeks
* Gastrointestinal endoscopy within the last 4 weeks
* Major gastrointestinal surgery (total/segmental gastrectomy, small bowel and/or colonic resection)
* Cholecystectomy
* Inflammatory bowel diseases
* Celiac disease
* Any etiology of chronic constipation other than FC (irritable bowel syndrome, rectocele, dyssynergic defecation, opioid use)
* Endocrine, metabolic or neurologic disorders causing constipation (hypothyroidism, Parkinson's disease, paraplegia)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Three or more complete bowel movements per week at 10 weeks | 10 weeks
  The proportion of patients with a mean of three or more complete bowel movements per week (CBMpW) at 10 weeks is compared between control and study groups.
Improvement in Patient Assessment Constipation Quality of Life | 10 weeks
  The proportion of the patients with more than 50% improvement in total Patient Assessment Constipation Quality of Life score is compared between control and study groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University Esenler Hospital, Istanbul, Other (Non U.s.), Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided